CLINICAL TRIAL: NCT03940079
Title: Efficacy of Computer-Based Cognitive Game Training on Motor and Cognitive Functions for Healthy Elderly
Brief Title: Efficacy of Computer-Based Cognitive Game Training for Healthy Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201804055RINC
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Aging; Cognitive Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gross-motor group (GMG) (Experimental): The participants of GMG received motor-cognitive dual-task training. The sensors used by the participants were four different colored buttons. The participants wear a suit with two buttons on the shoulders and the other two fasten on the knees by velcros. To accomplish the tasks, the participants had to slap the correct colored buttons. The stretching of upper or lower limbs was demanding while slapping, so the participants of GMG received a training which required cognitive and motor functions at the same time.
  The participants attended 2 sessions per week and lasted for 4 weeks. Each session lasted 75 minutes, mainly including 30 minutes for game introduction and warm-up, 30 minutes for game training, and 15 minutes for rest during the training. Each task lasted 10 minutes, and each session contained 3 tasks. The game difficulty could be adjusted automatically according to the performance of participants.
  Interventions: Device: computer-based cognitive game (including 3 training tasks)
- fine-motor group (FMG) (Active Comparator): The participants of FMG received cognitive training only. Four colored sensors used by the participants were the keys on the keyboard of the laptop. The participants simply pressed correct colored keys by fingers to complete the tasks.
  The participants attended 2 sessions per week and lasted for 4 weeks. Each session lasted 75 minutes, mainly including 30 minutes for game introduction and warm-up, 30 minutes for game training, and 15 minutes for rest during the training. Each task lasted 10 minutes, and each session contained 3 tasks. The game difficulty could be adjusted automatically according to the performance of participants.
  Interventions: Device: computer-based cognitive game (including 3 training tasks)

INTERVENTIONS:
Device: computer-based cognitive game (including 3 training tasks) — First task was short-term memory training. Participants were instructed to memorize different colored circles with ordinal numbers which would disappear later. They triggered correct colored sensor in sequence according to their memory.
  Second task was divided attention training. Different colored circles with ordinal numbers would not disappear this time.The participants should trigger correct colored sensor according to their sequence.
  Third task was inhibitory function training. There were red and green lights, just like the traffic light, hung up at the upper left of the scene. Red light represented prohibition of triggering the colored sensor, while green light urged to trigger it. Yellow, red, blue and green circles showed up randomly and moved toward the beige region. When the circle came extremely closer to the beige region, the traffic light was randomized to lighten up red or green.The participants should judge and trigger the correct colored sensor.

SUMMARY:
The declination on cognitive and motor functions in older adults increases the difficulty to achieve successful aging. Previous studies had reported that contrast to the traditional cognitive training methods, computer cognitive training (CCT) is comparable or has better effect on the cognitive function improvement with elders.On the other hand, some researchers claimed motor-cognitive dual-task training may possess greater effects than single cognitive training on cognitive functions. However, it is still on debate. Therefore, the research aims to investigate cognitive and motor benefits to healthy older adults over 65s trained by our computer-based cognitive game with high and low level of motor engagements.The research questions include: (1) Is CCT beneficial of cognitive functions? (2) Does CCT with high level of motor engagements (i.e. motor-cognitive dual-task training) have greater effects than single cognitive training on cognitive functions? (3) Can the training effect remain?

DETAILED DESCRIPTION:
Quasi-experimental design was adapted in our research.There are four time-series assessments during the experiment: baseline, pretest, posttest, and follow-up. After the baseline assessment, participants were randomized to two groups: gross-motor group (GMG) and fine-motor group (FMG). The intervals between baseline and pretest as well as between pretest and posttest were both 4 weeks, while the interval between posttest and follow-up was 8 weeks.

The investigators developed a computer-based cognitive game and compared the efficacy of cognitive and motor functions between computer-based cognitive game combining two different demands on motor control. Investigators hypothesized: All participants who take part in the computer-based cognitive game training don't have learning effects on pretest and are able to improve cognitive functions including short-term memory, divided attention and inhibitory function after intervention; Gross-motor group make more progress than fine-motor group on cognitive and motor functions after intervention. Furthermore, gross-motor group maintained more training effect over cognitive and motor functions at follow-up than fine-motor group.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 65 years old
2. Montreal Cognitive Assessment (MoCA) score ≥ 18
3. clear eyesight and hearing
4. both upper and lower limbs are functional
5. normal communication

Exclusion Criteria:

1. injury, fracture, and breathing problem
2. surgery during the research
3. severe disease affecting cognitive functions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Montreal Cognitive Assessment (MoCA) Taiwan Version at the 4th, 8th and 16th weeks | baseline, 4th weeks pretest, 8th weeks posttest, 16th weeks follow-up
  overall cognitive function
Change from Baseline Digit Span Task-forward (DS-forward) at the 4th, 8th and 16th weeks | baseline, 4th weeks pretest, 8th weeks posttest, 16th weeks follow-up
  short-term memory
Change from Baseline Color Trails Test-2 (CTT-2) at the 4th, 8th and 16th weeks | baseline, 4th weeks pretest, 8th weeks posttest, 16th weeks follow-up
  divided attention
Change from Baseline Stroop Color Word Test (SCWT) at the 4th, 8th and 16th weeks | baseline, 4th weeks pretest, 8th weeks posttest, 16th weeks follow-up
  inhibitory function
Change from Baseline Nine Hole Peg Test (NHPT) at the 4th, 8th and 16th weeks | baseline, 4th weeks pretest, 8th weeks posttest, 16th weeks follow-up
  motor function of upper limbs
Change from Baseline Get-Up and Go Test (GUG) at the 4th, 8th and 16th weeks | baseline, 4th weeks pretest, 8th weeks posttest, 16th weeks follow-up
  motor function of lower limbs and balance
Change from Baseline Five-Times-Sit-to-Stand Test (FTSST) at the 4th, 8th and 16th weeks | baseline, 4th weeks pretest, 8th weeks posttest, 16th weeks follow-up
  motor function of lower limbs and balance

SECONDARY OUTCOMES:
Change from 4th weeks Game1 (first scenario) evaluated the performance of short-term memory at 8th weeks | 4th weeks pretest, 8th weeks posttest
  Game assessment was a new way to evaluate cognitive performance of the participant through the score. All participants proceeded all three scenarios but challenged same degree of difficulty.
Change from 4th weeks Game2 (second scenario) evaluated divided attention at 8th weeks | 4th weeks pretest, 8th weeks posttest
  Game assessment was a new way to evaluate cognitive performance of the participant through the score. All participants proceeded all three scenarios but challenged same degree of difficulty.
Change from 4th weeks Game3 (third scenario) evaluated inhibitory function at 8th weeks | 4th weeks pretest, 8th weeks posttest
  Game assessment was a new way to evaluate cognitive performance of the participant through the score. All participants proceeded all three scenarios but challenged same degree of difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact Backup Mao, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No